CLINICAL TRIAL: NCT05551026
Title: Effects of Perioperative Operating Room Environment on Postoperative Delirium in Elderly Patients With Abdominal Surgery : A Prospective Cohort Study
Brief Title: Effects of Perioperative Operating Room Environment on Postoperative Delirium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Factors of POD
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thi investigators aims to observe the impact of perioperative body temperature and the noise of operating room on postoperative delirium for elderly patients undergoing abdominal surgery. And based on this study the investigators aimed to explore the potential risk factors of postoperative delirium for elderly patients undergoing abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-90 years old;
* ASA I-III;
* Patients who plan to undergo elective abdominal surgery under general anesthesia;
* Volunteer to participate in this study and sign informed consent.

Exclusion Criteria:

* Patients with known mental illness or lack of communication or cognitive impairment before operation;
* Severe vision, hearing, language impairment or other reasons unable to communicate with visitors;
* Severe dysfunction of important organs such as heart, brain, lung, liver, kidney, etc.;
* Long-term use of sedatives, antidepressants or alcoholism;
* Patients with severe postoperative complications and admitted to intensive care unit;
* Patients who refused or failed to complete the cognitive function test.
* Patients who could not cooperate with the study for any other reason.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients who underwent abdominal surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-26 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium during the 3 days-follow-up after anesthetic resuscitation | From ending of the surgery to 3 days after anesthetic resuscitation
  Postoperative delirium was tested with 3 minutes-Confusion Assessment Method or Confusion Assessment Method-intensive care unit (0-4, higher scores means worse outcome). The patient is determined to be postoperative delirium (ie, Confusion Assessment Method positive) if he/she fall ill quickly with confusion disorder, and with mental disorder or consciousness disorder.

SECONDARY OUTCOMES:
Postoperative delirium in the postanesthesia care unit | From ending of the surgery to the time when discharge from postanesthesia care unit, an average of 30 minutes
  Postoperative delirium was tested with 3 minutes-Confusion Assessment Method (0-4, higher scores means worse outcome). The patient is determined to be postoperative delirium (ie, Confusion Assessment Method positive) if he/she fall ill quickly with confusion disorder, and with mental disorder or consciousness disorder.
Hospital stay | From the ending of the surgery to hospital discharge, with means of about 7 days
  Time duration of the patients' stay in hospital
Postoperative complication | From the ending of the surgery to hospital discharge, with means of about 7 days
  The number of patients who having complication during the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jia Tang, MD, Study Director — Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China